CLINICAL TRIAL: NCT06349837
Title: Safety and Tolerability of Low Dose Radiotherapy Plus Concurrent Partial Stereotactic Ablative Radiotherapy (Eclipse-RT) and Tislelizumab in Patients With Bulky Tumors
Brief Title: Safety and Tolerability of LDRT Plus Concurrent Partial SBRT and Tislelizumab in Patients With Bulky Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, You Lu, Chair of Department of Thoracic Cancer, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECLIPSE-02
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor
Keywords: Low Dose Radiotherapy; Stereotactic Ablative Radiotherapy; Tislelizumab
MeSH Terms: interventions — tislelizumab; Immune Checkpoint Inhibitors; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDRT+SBRT + Tislelizumab (Experimental): This is a dose escalation study, low Dose Radiotherapy (LDRT) dose was 6Gy/3f, Stereotactic Ablative Radiotherapy (SBRT) dose was 24Gy/3f , 30Gy/3f and 45 Gy/3f, the dose of Tislelizumab was recommended in the instruction manual.
  Interventions: Drug: Tislelizumab; Radiation: Low Dose Radiotherapy; Radiation: Stereotactic Ablative Radiotherapy

INTERVENTIONS:
Drug: Tislelizumab — Patients will receive treatment with Tislelizumab (200 mg, iv, d1), every 3 weeks for a maximum of 48 months.
  Other Names: PD-1 inhibitor
Radiation: Low Dose Radiotherapy — LDRT (d1-d3): 6Gy/3f with conventional external beam radiation.
  Other Names: LDRT
Radiation: Stereotactic Ablative Radiotherapy — Partial SBRT at dose escalation levels: 24Gy/3f, 30Gy/3f, 45Gy/3f.
  Other Names: SBRT

SUMMARY:
This is a 3+3 dose escalation phase I study which aims to evaluate the safety and tolerability of low dose radiotherapy (LDRT) plus concurrent partial Stereotactic Ablative Radiotherapy (SBRT) and Tislelizumab in Patients with bulky tumors who have failed standard therapy. At least 9 participants will be enrolled in this study.

DETAILED DESCRIPTION:
This is 3+3 escalation phase I study which will be conducted in West China Hospital.

Step A: A dose escalation of low dose radiotherapy (LDRT) and partial SBRT, at least 3 patients per cohort (a total of at least 9 patients) will be enrolled to determine the maximum tolerated dose (MTD), dose-limiting toxicity (DLT) and recommended dose for expansion (RDE) for lung LDRT and partial SBRT.

All eligible patients will receive LDRT + partial SBRT and Tislelizumab at different dose levels (described as below). Tislelizumab will be given at 200mg as recommended in the instruction manual every 3 weeks until disease progression, unacceptable toxicities, the patient withdraws informed consent, or Tislelizumab reaches a maximum of up to 24 months.

Patients in the dose escalation will receive LDRT + partial SBRT at 3 cohorts with increasing dose levels: 6 Gy (2 Gy/f) + 24 Gy (8 Gy/f); 6 Gy (2 Gy/f) + 30 Gy (10 Gy/f); 6 Gy (2 Gy/f) + 45 Gy (15 Gy/f).

Step B: A dose expansion of LDRT + partial SBRT A cohort of 15 patients will receive lung LDRT and partial SBRT at the RDE determined during the dose-escalation phase in combination with PD-1 inhibitors to obtain additional safety and response data.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be ≥18 years of age on day of signing informed consent.
3. Patients with histologically or cytologically confirmed stage IV solid tumours.
4. Be willing to undergo repeat biopsy of tumor lesions according to the study protocol.
5. Patients who have failed the standard therapy, or who are unsuitable for standard treatment, or refuse chemotherapy.
6. At least one measurable lesion according to RECIST 1.1. A lesion that has previously received radiotherapy can be considered a target lesion only if this lesion is clearly progressed after radiotherapy.
7. The target lesions (irradiated lesions) are > 5cm in in diameter
8. ECOG 0-2.
9. Life expectancy of > 3 months.
10. Subjects should agree to use an adequate method of contraception.

Exclusion Criteria:

1. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis and/or spinal cord compression, etc.
2. With oncologic emergencies that require immediate treatment
3. EGFR/ALK/ROS-1 mutation or mutation status unknown.
4. Has evidence of interstitial lung disease or active and/or non-infectious pneumonitis (drug-induced pneumonia, radiation-induced pneumonia, etc.) requiring steroid therapy.
5. History of pulmonary fibrosis, pulmonary hypertension, severe irreversible airway obstruction disease
6. Patients with peripheral neuropathy.
7. Significant heart disease or impairment of cardiac function
8. Fluid accumulating in the third space, such as pericardial effusion, pleural effusion and peritoneal effusion that remains uncontrolled by aspiration or other treatment
9. Known allergy to drugs or excipients, known severe allergic reaction to any of the PD-1 monoclonal antibodies
10. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | 24 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months after the enrollment
  The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1.
Progression Free Survival (PFS) | up to 24 months after the enrollment
  Investigator assessed PFS according to RECIST v1.1. Progression free survival is defined as time of enrollment to first evidence of progressive disease.
Overall Survival (OS) | up to 24 months after the enrollment
  OS is defined as the difference (in months) between the date of study enrollment to the date death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yin L, Xue J, Li R, Zhou L, Deng L, Chen L, Zhang Y, Li Y, Zhang X, Xiu W, Tong R, Gong Y, Huang M, Xu Y, Zhu J, Yu M, Li M, Lan J, Wang J, Mo X, Wei Y, Niedermann G, Lu Y. Effect of Low-Dose Radiation Therapy on Abscopal Responses to Hypofractionated Radiation Therapy and Anti-PD1 in Mice and Patients With Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2020 Sep 1;108(1):212-224. doi: 10.1016/j.ijrobp.2020.05.002. Epub 2020 May 15. PMID 32417411
- [Background] Lan J, Li R, Yin LM, Deng L, Gui J, Chen BQ, Zhou L, Meng MB, Huang QR, Mo XM, Wei YQ, Lu B, Dicker A, Xue JX, Lu Y. Targeting Myeloid-derived Suppressor Cells and Programmed Death Ligand 1 Confers Therapeutic Advantage of Ablative Hypofractionated Radiation Therapy Compared With Conventional Fractionated Radiation Therapy. Int J Radiat Oncol Biol Phys. 2018 May 1;101(1):74-87. doi: 10.1016/j.ijrobp.2018.01.071. Epub 2018 Mar 12. PMID 29619980
- [Background] Zhou X, Zhou L, Yao Z, Huang M, Gong Y, Zou B, Zhu J, Liu Y, Peng F, Zhang Y, Yu M, Li Y, Na F, Wu Y, Kang K, Xiu W, Zhang X, Zhou L, Xu Y, Wang J, Wang Y, Yang X, Wu Y, Li R, Zhang Y, Yang Z, Zhou Z, Bai J, Yi X, Tong R, Yin L, Chen C, Niedermann G, Lu Y, Xue J. Safety and Tolerability of Low-Dose Radiation and Stereotactic Body Radiotherapy + Sintilimab for Treatment-Naive Stage IV PD-L1+ Non-Small Cell Lung Cancer Patients. Clin Cancer Res. 2023 Oct 13;29(20):4098-4108. doi: 10.1158/1078-0432.CCR-23-0315. PMID 37581611
- [Background] Zhou L, Liu Y, Wu Y, Yang X, Spring Kong FM, Lu Y, Xue J. Low-dose radiation therapy mobilizes antitumor immunity: New findings and future perspectives. Int J Cancer. 2024 Apr 1;154(7):1143-1157. doi: 10.1002/ijc.34801. Epub 2023 Dec 7. PMID 38059788
- [Background] Barsoumian HB, Ramapriyan R, Younes AI, Caetano MS, Menon H, Comeaux NI, Cushman TR, Schoenhals JE, Cadena AP, Reilly TP, Chen D, Masrorpour F, Li A, Hong DS, Diab A, Nguyen QN, Glitza I, Ferrarotto R, Chun SG, Cortez MA, Welsh J. Low-dose radiation treatment enhances systemic antitumor immune responses by overcoming the inhibitory stroma. J Immunother Cancer. 2020 Oct;8(2):e000537. doi: 10.1136/jitc-2020-000537. PMID 33106386
- [Background] Barsoumian HB, Sezen D, Menon H, Younes AI, Hu Y, He K, Puebla-Osorio N, Wasley M, Hsu E, Patel RR, Yang L, Cortez MA, Welsh JW. High Plus Low Dose Radiation Strategy in Combination with TIGIT and PD1 Blockade to Promote Systemic Antitumor Responses. Cancers (Basel). 2022 Jan 3;14(1):221. doi: 10.3390/cancers14010221. PMID 35008385
- [Background] Menon H, Chen D, Ramapriyan R, Verma V, Barsoumian HB, Cushman TR, Younes AI, Cortez MA, Erasmus JJ, de Groot P, Carter BW, Hong DS, Glitza IC, Ferrarotto R, Altan M, Diab A, Chun SG, Heymach JV, Tang C, Nguyen QN, Welsh JW. Influence of low-dose radiation on abscopal responses in patients receiving high-dose radiation and immunotherapy. J Immunother Cancer. 2019 Sep 4;7(1):237. doi: 10.1186/s40425-019-0718-6. PMID 31484556
- [Background] Welsh JW, Tang C, de Groot P, Naing A, Hess KR, Heymach JV, Papadimitrakopoulou VA, Cushman TR, Subbiah V, Chang JY, Simon GR, Ramapriyan R, Barsoumian HB, Menon H, Cortez MA, Massarelli E, Nguyen Q, Sharma P, Allison JP, Diab A, Verma V, Raju U, Shaaban SG, Dadu R, Cabanillas ME, Wang K, Anderson C, Gomez DR, Hahn S, Komaki R, Hong DS. Phase II Trial of Ipilimumab with Stereotactic Radiation Therapy for Metastatic Disease: Outcomes, Toxicities, and Low-Dose Radiation-Related Abscopal Responses. Cancer Immunol Res. 2019 Dec;7(12):1903-1909. doi: 10.1158/2326-6066.CIR-18-0793. Epub 2019 Oct 28. PMID 31658994